CLINICAL TRIAL: NCT00946959
Title: Characterization of Factors Influencing the Occurrence of Cognitive Decline in Patients With Coronary Artery Disease and Undergoing Cardiac Surgery and Coronary Angioplasty
Brief Title: Characterization of Factors Influencing the Cognitive Decline in Patients With Coronary Artery Disease
Acronym: COGCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2007_0724; 2007-A1420-53 (Other: ID-RCB Number, ANSM)
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
Keywords: cardiac surgery; angioplasty; cognitive decline
MeSH Terms: conditions — Coronary Artery Disease; Cognitive Dysfunction | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cardiac surgery (Experimental): This arm will include patients older than 18 years and candidate to cardiac surgery.
  Interventions: Procedure: Cardiac surgery
- cardiac angiography (No Intervention): Patients older than 18 years who undergo coronary angiogram. This arm will include patients with coronary revascularization and patients without coronary revascularization.

INTERVENTIONS:
Procedure: Cardiac surgery — A study-certified cardiothoracic surgeon must deem a patient, who otherwise fulfills all inclusion and exclusion criteria for any cardiac surgery (conventional, off-pump cardiac surgery). The procedure must be performed as soon as possible.
  Arms: cardiac surgery

SUMMARY:
The real impact of cardiac surgery and coronary angioplasty remains to be clarified and, where appropriate, the influencing factors in a way beneficial or deleterious remain to be identified.

The identification of such factors could make even faster screening, prevention and therefore open therapeutic prospects for those patients.

The objective of the study is to constitute a prospective cohort to assess the occurrence of cognitive decline after cardiac surgery (200 patients) and coronary angioplasty (200 patients) using the scale Dementia rating scale (DRS) of Mattis. In addition, the investigators will identify factors that influence positively or negatively, the occurrence of such a cognitive decline. The study based on a systematic monitoring of clinical, biological, imaging and pharmacological factors and, to correlate the respective influence of these factors on the incidence of cognitive decline.

DETAILED DESCRIPTION:
Cardiovascular invasive interventions (surgery and angioplasty) save thousands of lives every year, but questions remain about the neurological complications and in particular cognitive deficit. Indeed, cardiac surgery has been associated with cognitive decline in 50 to 70% of patients in the first postoperative week and in 20 to 40% of patients 6 months to one year after surgery.

The study will be based on a prospective monitoring during 1 year of a cohort of 400 patients who will receive either a cardiac surgery or coronary angioplasty. At inclusion, will be collected medical history, risk factors, treatment history, clinical and etiological data (imaging, cardiac and vascular balance).

The results of routine tests performed complementary to hospitalization will be recorded (echo-doppler vessels of the neck, cardiac ultrasound trans-thoracic and/or transesophageal a holter cardiac).

In recruiting, we will apply a method of matching based on age (on 5 years) between 2 groups in order to compare 2 homogeneous groups.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years,
* candidate to cardiac surgery or patients candidate to coronary angioplasty.

Exclusion Criteria:

* presenting a psychiatric illness that can interfere with the mental state and with scores provided in this study (explored in a systematic manner by the Mini International Neuropsychiatric Interview DSM 4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compare cognitive disorders using the scale Dementia rating scale (DRS) of Mattis in 2 groups | Before intervention and 12 month after intervention

SECONDARY OUTCOMES:
Blood biomarkers: inflammation, coagulation, protein | Before intervention, 3 weeks (no biology), 6 months (no MRI and biology) and 12 month after intervention (no biology)
Neuropsychological evaluation: global cognitive function using MMSE, memory, attention | Before intervention, 3 weeks (no biology), 6 months (no MRI and biology) and 12 month after intervention (no biology)
Imaging parameters (MRI): abnormalities of white matter, ischemic lesions, hippocampus volume | Before intervention, 3 weeks (no biology), 6 months (no MRI and biology) and 12 month after intervention (no biology)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Modine, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Cardiologique, CHRU de Lille, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No